CLINICAL TRIAL: NCT05698394
Title: Effect of Intravenous Low-dose Esketamine on Maternal Depression at 3 Years After Childbirth in Women With Prenatal Depression: 3-year Follow-up of a Randomized Controlled Trial
Brief Title: Effect of Low-dose Esketamine on Maternal Depression at 3 Years After Childbirth
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, MD, PHD, Professor and Chairman, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-562
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Prenatal Depression; Ketamine; Postpartum Depression
Keywords: Prenatal Depression; Esketamine; Postpartum Depression; Long-Term Prognosis
MeSH Terms: conditions — Depression, Postpartum | interventions — Esketamine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine group (Experimental): For women in this group, study drug (esketamine 0.2 mg/kg in 20 ml normal saline) will be infused at a rate of 30 ml/h (infusion finished in 40 minutes) after giving birth.
  Interventions: Drug: Esketamine
- placebo group (Placebo Comparator): For women in this group, study drug (20 ml normal saline) will be infused at a rate of 30 ml/h (infusion finished in 40 minutes) after giving birth.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esketamine — 0.2 mg/kg S-ketamine in 20 ml normal saline will be infused at a rate of 30 ml/h (infusion finished in 40 minutes) after giving birth
  Arms: Esketamine group
Drug: Placebo — 20 ml normal saline will be infused at a rate of 30 ml/h (infusion finished in 40 minutes) after giving birth.
  Other Names: normal saline; 0.9% sodium chloride
  Arms: placebo group

SUMMARY:
Postpartum depression refers to the depression after childbirth, which is a common mental disorder in women. The pathogenesis of postpartum depression is not fully understood, and may be related to a variety of factors. Prenatal depression is an important risk factor for postpartum depression. Our recent multicenter randomized controlled trial, "Effect of Low-dose esketamine on the incidence of postpartum depression in women with prenatal depression", explored the effect of immediate postpartum intravenous infusion of low-dose esketamine on the incidence of postpartum depression in women with prenatal depression. The preliminary results showed that it reduced the incidence of postpartum depression at 42 days. Since there were no studies on the effect of intravenous esketamine infusion after delivery on long-term postpartum depression, this study is a long-term follow-up of the previous randomized trial. We aim to explore the effect of low-dose intravenous esketamine after delivery on the incidence of 2-year maternal depression after delivery in women with prenatal depressive symptoms.

DETAILED DESCRIPTION:
Postpartum depression refers to the depression after childbirth. It is a common mental disorder after childbirth. In recent years, it has attracted more and more public attention. Studies have reported an incidence of postpartum depression ranging from 10% to 29%. Our previous findings showed that the incidence of depression at 42 days postpartum was 24.3%. Postpartum depression has adverse effects on physical and mental health of women, but also may have adverse influences on offspring including nutrition health, and cognitive and behavioral development. The pathogenesis of postpartum depression is not completely clear, and may be related to many factors, such as hormone level changes after childbirth, psychosocial factors, and adverse obstetric factors. Plently of studies have shown that prenatal depression is an important risk factor for postpartum depression. One meta-analysis showed that the incidence of postnatal depression could be as high as 39% in people with prenatal depression. Therefore, it is possible to reduce the occurrence of postpartum depression by active intervention of prenatal depressed parturients.

Ketamine, an NMDA-receptor antagonist, is a classic analgesic drug with advantages of light respiratory and circulatory inhibition and good analgesic effect. Recently, it has been found to have antidepressant effect and has been widely used in the field of psychiatry. Esketamine, a S-enantiomer of racemic ketamine, has similar antidepressant effects to equivalent doses of ketamine, with a lower incidence of adverse reactions. In 2019, esketamine was approved by the US FDA for the treatment of treatment-resistant depression. At present, the results of studies on the use of esketamine in the perioperative period for the prevention and treatment of postoperative or postpartum depression are mixed.

Our recent multicenter randomized controlled trial, "Effect of low-dose esketamine on the incidence of postpartum depression in women with prenatal depression", explored the effect of immediate postpartum intravenous administration of low-dose esketamine on the incidence of postpartum depression in women with prenatal depression. The multicenter study included 364 women who were given a low dose of esketamine intravenously after delivery. Preliminary results show that it can reduce the incidence of postpartum depression at 42 days. Here we conduct a 2-year follow-up of the women enrolled in the underlying trial to figure out the occurrence of 2-year maternal depression, and to explore the effect of immediate intravenous infusion of low-dose esketamine on the incidence of chronic depression at 2 years postpartum.

ELIGIBILITY:
All 364 pregnant women who participated in the underling trial "Effect of low-dose esketamine on the incidence of postpartum depression in women with prenatal depression: a randomized, double-blind, placebo-controlled trial" NCT04414943）and agreed to accept this 2-year follow-up.

The inclusion criteria of the underlying trial:

* Maternal age ≥18 years;
* Prenatal Edinburgh postnatal depression scale score ≥10 points.

Exclusion Criteria of the previous study:

* A clear history of mental illness (depression, schizophrenia, etc.) or communication disorders
* Severe pregnancy complications (such as severe preeclampsia, placenta accreta, HELLP syndrome, placenta previa, placenta abruption) before surgery;
* ASA grade ≥III;
* The presence of contraindications to ketamine/esketamine use (e.g., stubborn, refractory hypertension, severe cardiovascular disease [cardiac function grade ≥III], hyperthyroidism).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 364 (Actual)
Dates: Start 2023-09-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Incidence maternal depression at 3 years postpartum | At 3 years postpartum (33-41 months)
  Incidence of depression in women at 3 years postpartum. Diagnosis was made according to M.I.N.I. 6.0.

SECONDARY OUTCOMES:
PHQ-9 scores and incidence of moderate-severe depression in women at 3 years postpartum. | At 3 years postpartum (33-41 months)
  PHQ-9 score and moderate-severe depression (PHQ-9 score ≥10) in women at 3 years postpartum.
Incidence of chronic pain in women at 3 years postpartum | At 3 years postpartum (33-41 months)
  Incidence of chronic pain in women at 3 years postpartum
Incidence of developmental delay in offspring at 3 years of age | At 3 years postpartum (33-41 months)
  Incidence of developmental delay in offspring at 3 years of age measured by the Ages & Stages Questionnaires 3rd edition (ASQ-3) in Chinese

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (4):
- China (4):
  - Hunan Provincial Maternal and Child Health Care Hospital, Changsha, Hunan
  - Women's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Women's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woody CA, Ferrari AJ, Siskind DJ, Whiteford HA, Harris MG. A systematic review and meta-regression of the prevalence and incidence of perinatal depression. J Affect Disord. 2017 Sep;219:86-92. doi: 10.1016/j.jad.2017.05.003. Epub 2017 May 8. PMID 28531848
- [Background] Stewart DE, Vigod SN. Postpartum Depression: Pathophysiology, Treatment, and Emerging Therapeutics. Annu Rev Med. 2019 Jan 27;70:183-196. doi: 10.1146/annurev-med-041217-011106. PMID 30691372
- [Background] Deng CM, Ding T, Li S, Lei B, Xu MJ, Wang L, Xu SC, Yang HX, Sun XY, Li XY, Ma D, Wang DX. Neuraxial labor analgesia is associated with a reduced risk of postpartum depression: A multicenter prospective cohort study with propensity score matching. J Affect Disord. 2021 Feb 15;281:342-350. doi: 10.1016/j.jad.2020.12.027. Epub 2020 Dec 8. PMID 33348177
- [Background] O'Hara MW, McCabe JE. Postpartum depression: current status and future directions. Annu Rev Clin Psychol. 2013;9:379-407. doi: 10.1146/annurev-clinpsy-050212-185612. Epub 2013 Feb 1. PMID 23394227
- [Background] Stein A, Pearson RM, Goodman SH, Rapa E, Rahman A, McCallum M, Howard LM, Pariante CM. Effects of perinatal mental disorders on the fetus and child. Lancet. 2014 Nov 15;384(9956):1800-19. doi: 10.1016/S0140-6736(14)61277-0. Epub 2014 Nov 14. PMID 25455250
- [Background] Aoyagi SS, Tsuchiya KJ. Does maternal postpartum depression affect children's developmental outcomes? J Obstet Gynaecol Res. 2019 Sep;45(9):1809-1820. doi: 10.1111/jog.14064. Epub 2019 Jul 18. PMID 31321836
- [Background] Pearlstein T, Howard M, Salisbury A, Zlotnick C. Postpartum depression. Am J Obstet Gynecol. 2009 Apr;200(4):357-64. doi: 10.1016/j.ajog.2008.11.033. PMID 19318144
- [Background] Underwood L, Waldie K, D'Souza S, Peterson ER, Morton S. A review of longitudinal studies on antenatal and postnatal depression. Arch Womens Ment Health. 2016 Oct;19(5):711-20. doi: 10.1007/s00737-016-0629-1. Epub 2016 Apr 16. PMID 27085795
- [Background] Duman RS, Aghajanian GK. Synaptic dysfunction in depression: potential therapeutic targets. Science. 2012 Oct 5;338(6103):68-72. doi: 10.1126/science.1222939. PMID 23042884
- [Background] McIntyre RS, Rosenblat JD, Nemeroff CB, Sanacora G, Murrough JW, Berk M, Brietzke E, Dodd S, Gorwood P, Ho R, Iosifescu DV, Lopez Jaramillo C, Kasper S, Kratiuk K, Lee JG, Lee Y, Lui LMW, Mansur RB, Papakostas GI, Subramaniapillai M, Thase M, Vieta E, Young AH, Zarate CA Jr, Stahl S. Synthesizing the Evidence for Ketamine and Esketamine in Treatment-Resistant Depression: An International Expert Opinion on the Available Evidence and Implementation. Am J Psychiatry. 2021 May 1;178(5):383-399. doi: 10.1176/appi.ajp.2020.20081251. Epub 2021 Mar 17. PMID 33726522
- [Background] Correia-Melo FS, Leal GC, Vieira F, Jesus-Nunes AP, Mello RP, Magnavita G, Caliman-Fontes AT, Echegaray MVF, Bandeira ID, Silva SS, Cavalcanti DE, Araujo-de-Freitas L, Sarin LM, Tuena MA, Nakahira C, Sampaio AS, Del-Porto JA, Turecki G, Loo C, Lacerda ALT, Quarantini LC. Efficacy and safety of adjunctive therapy using esketamine or racemic ketamine for adult treatment-resistant depression: A randomized, double-blind, non-inferiority study. J Affect Disord. 2020 Mar 1;264:527-534. doi: 10.1016/j.jad.2019.11.086. Epub 2019 Nov 14. PMID 31786030
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Papakostas GI, Salloum NC, Hock RS, Jha MK, Murrough JW, Mathew SJ, Iosifescu DV, Fava M. Efficacy of Esketamine Augmentation in Major Depressive Disorder: A Meta-Analysis. J Clin Psychiatry. 2020 May 26;81(4):19r12889. doi: 10.4088/JCP.19r12889. PMID 32459407
- [Background] Singh JB, Daly EJ, Mathews M, Fedgchin M, Popova V, Hough D, Drevets WC. Approval of esketamine for treatment-resistant depression. Lancet Psychiatry. 2020 Mar;7(3):232-235. doi: 10.1016/S2215-0366(19)30533-4. No abstract available. PMID 32087801
- [Background] Pang L, Cui M, Dai W, Kong J, Chen H, Wu S. Can Intraoperative Low-Dose R,S-Ketamine Prevent Depressive Symptoms After Surgery? The First Meta-Analysis of Clinical Trials. Front Pharmacol. 2020 Oct 19;11:586104. doi: 10.3389/fphar.2020.586104. eCollection 2020. PMID 33192527
- [Background] Wang Q, Xiao M, Sun H, Zhang P. A Study on the Preventive Effect of Esketamine on Postpartum Depression (PPD) after Cesarean Section. Comput Math Methods Med. 2022 Aug 8;2022:1524198. doi: 10.1155/2022/1524198. eCollection 2022. PMID 35979054
- [Background] Wang Y, Zhang Q, Dai X, Xiao G, Luo H. Effect of low-dose esketamine on pain control and postpartum depression after cesarean section: a retrospective cohort study. Ann Palliat Med. 2022 Jan;11(1):45-57. doi: 10.21037/apm-21-3343. PMID 35144397
- [Background] Han Y, Li P, Miao M, Tao Y, Kang X, Zhang J. S-ketamine as an adjuvant in patient-controlled intravenous analgesia for preventing postpartum depression: a randomized controlled trial. BMC Anesthesiol. 2022 Feb 16;22(1):49. doi: 10.1186/s12871-022-01588-7. PMID 35172727
- [Background] Liu ZH, He ST, Deng CM, Ding T, Xu MJ, Wang L, Li XY, Wang DX. Neuraxial labour analgesia is associated with a reduced risk of maternal depression at 2 years after childbirth: A multicentre, prospective, longitudinal study. Eur J Anaesthesiol. 2019 Oct;36(10):745-754. doi: 10.1097/EJA.0000000000001058. PMID 31356375
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Wang W, Bian Q, Zhao Y, Li X, Wang W, Du J, Zhang G, Zhou Q, Zhao M. Reliability and validity of the Chinese version of the Patient Health Questionnaire (PHQ-9) in the general population. Gen Hosp Psychiatry. 2014 Sep-Oct;36(5):539-44. doi: 10.1016/j.genhosppsych.2014.05.021. Epub 2014 Jun 6. PMID 25023953